CLINICAL TRIAL: NCT01393158
Title: A Pilot Study of an Oral Phosphodiesterase Inhibitor (Apremilast) for Atopic Dermatitis in Adults
Brief Title: Apremilast for Atopic Dermatitis - A Pilot Study in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Eric Simpson, Associate Professor, Dermatology, Oregon Health and Science University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP-PI-AD-0034
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: 20mg cohort enrolled and completed before the 30mg cohort enrolled.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20 mg BID (Experimental): Patients dosed with 20 mg orally of Apremilast BID for 3 months.
  Interventions: Drug: Apremilast
- 30 mg BID (Experimental): Patients dosed with 30 mg orally of Apremilast BID for 6 months.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 20mg of Apremilast taken orally BID for 3 months or 30 mg of Apremilast taken orally BID for 6 months.
  Other Names: Otezla

SUMMARY:
The purpose of this study is to obtain preliminary data regarding the safety and tolerability of apremilast in AD to support the design of larger controlled studies.

DETAILED DESCRIPTION:
To investigate the preliminary safety and efficacy of apremilast, an oral phosphodiesterase 4 inhibitor, for atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Disease severity of Moderate, Severe, or Very Severe by Investigator Global Assessment.
* Disease severity must be greater than or equal to 6 on the Rajka-Langeland Severity Scoring system corresponding to moderate-severe disease.
* Baseline EASI score must be greater than or equal to 11. A previous validation study for the EASI scoring system revealed patients with moderate to very severe disease had mean EASI scores ranging from 11-30.
* Candidate for, or previously on systemic therapy, including cyclosporine, methotrexate, or other immunosuppressant and treatment with ultraviolet light. Specifically, subjects are considered candidates for systemic therapy when their disease is not adequately controlled using topical therapies or side-effects prevent the further safe use of topical therapies.
* Subjects must meet the washout requirements

Exclusion Criteria:

* History of active mycobacterial infection with any species (including Mycobacterium tuberculosis) within 3 years prior to screening visit. Subjects with Mycobacterium tuberculosis infection more than 3 years prior to screening visit are allowed if successful treatment was completed at least 3 years prior to randomization and is documented and available for verification.
* At least 3 major bacterial infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years.
* Clinically significant abnormality on the chest X-ray (CXR) at screening. Chest X-rays performed within 3 months prior to start of study drug are acceptable.
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer).
* Any clinically significant abnormality on 12-lead ECG (electrocardiogram) at screening.
* History of congenital or acquired immunodeficiency (e.g., Common Variable Immunodeficiency [CVID]).
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening.
* History of Human Immunodeficiency Virus (HIV) infection.
* Antibodies to Hepatitis C at screening.
* History of squamous cell carcinoma of the skin and thin melanoma.
* Systemic corticosteroid-dependent asthma.
* Active infection of any type at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Simpson, MD, MCR, Principal Investigator — Oregon Health and Science University

REFERENCES:
- [Derived] Samrao A, Berry TM, Goreshi R, Simpson EL. A pilot study of an oral phosphodiesterase inhibitor (apremilast) for atopic dermatitis in adults. Arch Dermatol. 2012 Aug;148(8):890-7. doi: 10.1001/archdermatol.2012.812. PMID 22508772

RESULTS

PARTICIPANT FLOW:
Groups:
- Apremilast 20mg: Apremilast: 20 mg by mouth twice daily for a total of 12 weeks.
- Apremilast 30mg: Apremilast: 30 mg by mouth twice daily for a total of 24 weeks.
Period: Overall Study
Arm/Group | Apremilast 20mg | Apremilast 30mg
Started | 6 | 10
Completed | 5 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apremilast 20mg | Apremilast 30mg | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 10 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
EASI [Mean (Standard Deviation); unit: units on a scale] — The eczema area and severity index (EASI) is a validated composite score measuring physical signs of atopic dermatitis. The scale ranges from 0-72. The components measuring severity are four symptoms of eczema: erythema, population, excoriation and lichenification on a scale of 0-3 for each body of the four body regions (head/neck, trunk, arms, legs). The score for each patient's with scores between 0 and 7 are considered mild ,between 7 and 21 are considered moderate, and greater than 21 are considered severe.
  units on a scale | 30.9 (12.0) | 21.4 (7.6) | 24.8 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in EASI Scores
Description: The eczema area and severity index (EASI) is a composite score measuring physical signs of atopic dermatitis. The scale ranges from 0-72. The components measuring severity are four signs/symptoms of atopic dermatitis: erythema, population, excoriation and lichenification on a scale of 0-3 for each body of the four body regions (head/neck, trunk, arms, legs). The component measuring area is a body surface area measurement of each region. The area and severity of each body region is weighted based on size of region which are added together for the complete score. The score for each patient's with scores between 0 and 7 are considered mild ,between 7 and 21 are considered moderate, and greater than 21 are considered severe. In this study the change in EASI score between baseline and month three (end of study) in the 20 mg arm and month six in the 30 mg arm, baseline EASI score was subtracted from month 3 or month 6 score in the 30mg arm,and calculated as a final outcome data point.
Time Frame: Mean change in EASI score measured at Baseline and Month 3, (if on 20mg arm) or Baseline and Month 6 (if on 30mg arm)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Apremilast 20 BID: Subjects received 20mg of Apremilast BID for 12 weeks
- Apremilast 30mg BID: Subjects received 30mg of Apremilast BID for 24 weeks
Arm/Group | Apremilast 20 BID | Apremilast 30mg BID
Number analyzed (Participants) | 6 | 10
units on a scale | -8.8 (11.6) | -8.2 (9.1)

2. Secondary Outcome: Number of Participants in Each IGA Category
Description: The investigator global assessment scale is a gestalt global assessment made by an investigator describing the overall disease severity of the patient. It is a categorical scale that includes 0-clear, 1-almost clear, 2-mild,3- moderate, 4-severe, and 5-very severe. The reduction in IGA score from baseline to month three (end of study) in the 20mg arm and month six (end of study) in the 30mg arm was evaluated for efficacy.
Time Frame: Mean change in IGA score measured at Baseline and Month 3, (if on 20mg arm) or Baseline and Month 6 (if on 30mg arm)
Measure: Number; unit: participants
Groups:
- Apremilast 20 BID: Subjects received 20mg BID for 12 weeks
- Apremilast 30 BID: Subjects received 30mg of Apremilast BID for 24 weeks
Arm/Group | Apremilast 20 BID | Apremilast 30 BID
Number analyzed (Participants) | 6 | 10
participants
  Mild | 0 | 1
  Moderate | 2 | 8
  Severe | 3 | 1
  Very Severe | 1 | 0

3. Secondary Outcome: Change in Pruritus (Visual Analog Scale) Score
Description: The pruritus visual analog scale (VAS) is a 10 cm (100 mm) visual analog scale that measures up patient's itch severity with 10 (100 mm) representing the worst imaginable and 0 representing no itch. This is a validated scale with a change of three from baseline to month three in the 20mg arm (end of study) and month six in the 30mg arm (end of study) being clinically relevant.
Time Frame: Mean change in Pruritus (Visual Analog Scale) score measured at Baseline and Month 3, (if on 20mg arm) or Baseline and Month 6 (if on 30mg arm)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Apremilast 20mg BID: Subjects received 20mg BID
- Apremilast 30mg BID: Subjects received 30 mg BID
Arm/Group | Apremilast 20mg BID | Apremilast 30mg BID
Number analyzed (Participants) | 6 | 10
units on a scale | -32.2 (24.0) | -13.4 (22.0)

4. Secondary Outcome: Change In DLQI Scores
Description: The dermatology life quality index (DLQI) is a validated quality-of-life scale that measures the impact of skin disease. It is a 10 question instrument. Scores of 0 over 0-1 means there is no effect on the patient's life. Scores between 2 and 5 represent a small effect on patient's life. Scores between 6 and 10 correspond to a moderate effect on patient's life. Scores between 11 and 20 correspond to a very large effect on the patient's life. And scores between 21 and 30 correspond to an extremely large effect on patient's life. The range of the scale between 0 and 30 for the added total of the patient's responses. Each question can be answered on a scale of 0-"not at all", 1-"a little", 2-" a lot", 3- "very much" with some questions having the option of "not relevant". The difference in DLQI score from baseline to month three (end of study) in the 20mg arm and month six (end of study) in the 30mg arm was evaluated for efficacy.
Time Frame: Mean change in DLQI scores measured at Baseline and Month 3, (if on 20mg arm) or Baseline and Month 6 (if on 30mg arm)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Apremilast 20 BID: Subjects received 20mg Apremilast BID
- Apremilast 30mg BID: Subjects received 30mg Apremilast BID
Arm/Group | Apremilast 20 BID | Apremilast 30mg BID
Number analyzed (Participants) | 6 | 10
units on a scale | -8.3 (4.0) | -6.3 (5.6)

ADVERSE EVENTS:
Time Frame: 4 Months in the 20 mg BID arm, and 7 months in the 30mg BID arm.
Description: All-cause mortality was not monitored/assessed.
Groups:
- Apremalist 20mg BID: Patients receiving 20mg BID for 12 weeks
- Apremalist 30mg BID: Patients receiving 30mg BID for 24 weeks
Arm/Group | Apremalist 20mg BID | Apremalist 30mg BID
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 2/6 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremalist 20mg BID (N=6) | Apremalist 30mg BID (N=10)
Nausea (Gastrointestinal disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No